CLINICAL TRIAL: NCT00787176
Title: The Association Between Fluid Administration, Oxytocin Administration, and Fetal Heart Rate Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study concluded prematurely prior to meeting intended goal recruitment.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Paloma Toledo, Associate Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0524-034
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy; Labor Pain
Keywords: Oxytocin; Labor, Obstetric; Non-reassuring fetal heart rate; epidural
MeSH Terms: conditions — Labor Pain | interventions — Ringer's Lactate; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient is positioned for epidural placement. Oxytocin management continued as per protocol.
  Interventions: Drug: Group A Intravenous bolus of 1000 ml lactated ringers solution
- Group B (Experimental): An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
  Interventions: Drug: Group B Intravenous bolus bolus 1000 ml lactated ringers solution oxytocin decrease to 1/2 current rate
- Group C (Active Comparator): The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
  Interventions: Drug: Group C 125 mL/hr of lactated ringers
- Group D (Experimental): The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement was halved and not increased for 60 minutes until after placement.
  Interventions: Drug: Group D 125 mL/hr lactated ringers oxytocin decreased to 1/2 current rate

INTERVENTIONS:
Drug: Group A Intravenous bolus of 1000 ml lactated ringers solution — An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient was positioned for epidural placement. Oxytocin management continued as per protocol.
  Other Names: A
  Arms: Group A
Drug: Group B Intravenous bolus bolus 1000 ml lactated ringers solution oxytocin decrease to 1/2 current rate — An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
  Other Names: B
  Arms: Group B
Drug: Group C 125 mL/hr of lactated ringers — The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
  Other Names: C
  Arms: Group C
Drug: Group D 125 mL/hr lactated ringers oxytocin decreased to 1/2 current rate — The maintenance infusion of 125 mL/hr of Lactated Ringers was given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
  Other Names: D
  Arms: Group D

SUMMARY:
Fetal heart rate patterns are an important parameter in the diagnosis of non-reassuring fetal status. Combined-spinal epidural analgesia is a method of initiating labor analgesia used by approximately 90% of the parturients at Prentice Women's Hospital. Optimizing the variables which could affect fetal heart rate patterns at the time of initiation of analgesia, such as fluid administration and oxytocin management, could help us provide better care for our patients and their fetuses.

Hypotheses: The combination of fluid administration and lower doses of oxytocin administration will have fewer adverse fetal heart rate changes in the first 60 minutes following initiation of labor analgesia.

DETAILED DESCRIPTION:
After obtaining informed, written consent, candidates were randomized to one of four groups at the time of request for labor analgesia. All subjects received a maintenance infusion of Lactated Ringers(LR). For candidates in Groups A or B, an intravenous bolus of 1000 mL of LR was initiated. Candidates in Groups C and D did not receive any additional fluid. If randomized to group A or C, the oxytocin management was continued as per the normal active management of labor protocal (AMOL). If randomized to groups B or D, the dose of oxytocin that was being administered was halved and not increased until 60 minutes after the initiation of epidural analgesia. Fetal heart rate monitoring and frequency of uterine contractions were recorded by external tocodynamometry.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Healthy nulliparous or multiparous women
* Term (>36 week gestation)
* Singleton pregnancy
* Spontaneous labor or with spontaneous rupture of membranes
* Receive oxytocin
* Request neuraxial analgesia

Exclusion Criteria:

* Under 18 years of age
* Presence of any systemic disease (e.g., diabetes mellitus, hypertension, preeclampsia)
* Use of chronic analgesic medications
* Prior administration of systemic opioid labor analgesia
* Non-vertex presentation
* Induction of labor
* Contraindication to neuraxial analgesia.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Toledo, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Prentice Women's Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mardirosoff C, Dumont L, Boulvain M, Tramer MR. Fetal bradycardia due to intrathecal opioids for labour analgesia: a systematic review. BJOG. 2002 Mar;109(3):274-81. doi: 10.1111/j.1471-0528.2002.01380.x. PMID 11950182
- [Background] Clarke VT, Smiley RM, Finster M. Uterine hyperactivity after intrathecal injection of fentanyl for analgesia during labor: a cause of fetal bradycardia? Anesthesiology. 1994 Oct;81(4):1083. doi: 10.1097/00000542-199410000-00041. No abstract available. PMID 7943823
- [Background] Lopez-Zeno JA, Peaceman AM, Adashek JA, Socol ML. A controlled trial of a program for the active management of labor. N Engl J Med. 1992 Feb 13;326(7):450-4. doi: 10.1056/NEJM199202133260705. PMID 1732771

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Full Oxytocin 1000 ml LR: An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient is positioned for epidural placement. Oxytocin management continued as per protocol.
  Group A: An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient was positioned for epidural placement. Oxytocin management continued as per protocol.
- Group B 1/2 Oxytocin 1000 ml LR: An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
  Group B: An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
- Group C Full Oxytocin No LR: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
  Group C: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
- Group D 1/2 Oxytocin no Additional LR: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement was halved and not increased for 60 minutes until after placement.
  Group D: The maintenance infusion of 125 mL/hr of Lactated Ringers was given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
Period: Overall Study
Arm/Group | Group A Full Oxytocin 1000 ml LR | Group B 1/2 Oxytocin 1000 ml LR | Group C Full Oxytocin No LR | Group D 1/2 Oxytocin no Additional LR
Started | 69 | 62 | 60 | 60
Completed | 62 | 59 | 54 | 55
Not Completed | 7 | 3 | 6 | 5
Not completed — Low quality fetal heart rate tracing | 7 | 3 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Group A: An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient is positioned for epidural placement. Oxytocin management continued as per protocol.
  Group A: An intravenous bolus of 1000 mL Lactated Ringers initiated when the patient was positioned for epidural placement. Oxytocin management continued as per protocol.
- Group B: An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
  Group B: An intravenous bolus of 1000 mL Lactated Ringers. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
- Group C: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
  Group C: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. Oxytocin management continued per protocol.
- Group D: The maintenance infusion of 125 mL/hr of Lactated Ringers will be given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement was halved and not increased for 60 minutes until after placement.
  Group D: The maintenance infusion of 125 mL/hr of Lactated Ringers was given with no additional fluid bolus. The dose of oxytocin being administered at time of epidural placement will be halved and not increased for 60 minutes until after placement.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 69 | 62 | 60 | 60 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 69 | 62 | 60 | 60 | 251
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.14 (4.97) | 30.50 (5.27) | 31.15 (4.34) | 30.42 (5.88) | 30.8 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 62 | 60 | 60 | 251
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 62 | 60 | 60 | 251
Region of Enrollment [Number; unit: participants] — Enrolled at Northwestern Medicine, Chicago,IL USA
  participants
    United States | 69 | 62 | 60 | 60 | 251
Body Mass Index (kg/m∧ 2) [Mean (Standard Deviation); unit: (kg/m∧ 2)] | 29.64 (4.49) | 28.26 (3.63) | 30.77 (6.1) | 30.51 (5.96) | 29.8 (5.05)
Estimated Gestational Age (weeks) [Mean (Standard Deviation); unit: Weeks] | 39.18 (1.17) | 39.06 (1.21) | 39.6 (1.04) | 39.02 (1.34) | 39.22 (1.19)
Baseline oxytocin (milliunit/minute) [Mean (Standard Deviation); unit: (milliunit/minute)] | 6.54 (4.64) | 6.65 (4.04) | 6.15 (5.16) | 5.88 (4.26) | 6.3 (4.5)
Cervical Dilation (cm) [Mean (Standard Deviation); unit: centimeters] | 3.54 (1.10) | 3.72 (1.01) | 3.6 (1.32) | 3.52 (1.01) | 3.6 (1.11)
Number of times pregnant [Number; unit: participants]
  1 pregnancy | 36 | 38 | 33 | 40 | 147
  2 pregnancies | 20 | 9 | 14 | 8 | 51
  3 pregnancies | 5 | 6 | 6 | 7 | 24
  4 pregnancies | 5 | 5 | 2 | 2 | 14
  5 pregnancies | 1 | 1 | 2 | 1 | 5
  6 pregnancies | 2 | 2 | 1 | 1 | 6
  7 pregnancies | 0 | 1 | 1 | 0 | 2
  8 pregnancies | 0 | 0 | 1 | 1 | 2
Number of live births [Number; unit: participants]
  0 live births | 49 | 44 | 42 | 47 | 182
  1 live birth | 14 | 13 | 12 | 10 | 49
  2 live births | 4 | 2 | 4 | 1 | 11
  3 live births | 2 | 2 | 1 | 1 | 6
  4 live births | 0 | 1 | 1 | 0 | 2
  5 live births | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-reassuring Fetal Heart Rate Tracings During the First 30 Minutes After the Placement of Epidural Analgesia
Description: The number of participants who experience non-reassuring fetal heart rate tracings obtained via electronic recording during the first 30 minutes after the placement of epidural analgesia
Time Frame: Request for labor analgesia up to the first 30 minutes after the placement of epidural
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 62 | 59 | 54 | 55
participants
  Favorable fetal heart rate tracings | 47 | 54 | 44 | 47
  Non reassuring fetal heart rate tracings | 15 | 5 | 10 | 8

2. Post Hoc Outcome: Delivery Type
Description: Type of delivery (vaginal, forceps assisted, cesarean, emergency cesarean section)
Time Frame: Delivery
Measure: Number; unit: participants
Groups:
- Group Sum: Sum of the four groups
Arm/Group | Group A | Group B | Group C | Group D | Group Sum
Number analyzed (Participants) | 69 | 62 | 60 | 60 | 251
participants
  Normal spontanous vaginal delivery | 50 | 43 | 44 | 44 | 181
  Forceps assisted vaginal delivery | 6 | 8 | 2 | 6 | 22
  Cesarean delivery | 13 | 11 | 14 | 10 | 48

ADVERSE EVENTS:
Time Frame: To time of delivery of baby.
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/62 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/62 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/69 | 0/62 | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=69) | Group B (N=62) | Group C (N=60) | Group D (N=60)
Cesarean Section for Fetal Distress (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Need for Cesarean delivery because of fetal distress or intolerance.

LIMITATIONS AND CAVEATS:
Study recruitment was stopped before reaching the determined a priori sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-06-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT00787176/Prot_SAP_000.pdf